CLINICAL TRIAL: NCT00729846
Title: Combination Bevacizumab and Verteporfin (Standard and Reduced Fluence)in the Treatment of Neovascular Age-Related Macular Degeneration
Brief Title: Bevacizumab in Combination With Visudyne Photodynamic Therapy (PDT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Dante Pieramici, Director of Research, California Retina Consultants
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPDT2006
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-03

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization; Macular Edema
Keywords: choroidal neovascularization; macular degeneration; macular edema; intravitreal bevacizumab; vegf; verteporfin PDT
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Macular Edema | interventions — Bevacizumab; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients will receive combination verteporfin with photodynamic therapy at reduced fluence [300mw/cm2] followed by intravitreal bevacizumab (1.25mg) on same day following photodynamic therapy.
  Interventions: Drug: Bevacizumab; Device: verteporfin photodynamic therapy reduced fluence
- B (Experimental): Patients will receive combination verteporfin with photodynamic therapy at standard fluence [600mw/cm2] followed by intravitreal bevacizumab (1.25mg) on same day following photodynamic therapy.
  Interventions: Drug: Bevacizumab; Device: verteporfin photodynamic therapy standardfluence

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive intravitreal bevacizumab (1.25mg) on same day following photodynamic therapy.
  Other Names: Avastin, visudyne
Device: verteporfin photodynamic therapy reduced fluence — Patients will receive combination verteporfin photodynamic therapy with stand fluence [600mW/cm2].
  Other Names: PDT
  Arms: A
Device: verteporfin photodynamic therapy standardfluence — Patients will receive combination verteporfin with photodynamic therapy at standard fluence [600mw/cm2].
  Arms: B

SUMMARY:
To evaluate safety, visual acuity outcomes, persistence of choroidal neovascular leakage, and the number of treatments of combination intravitreal bevacizumab and verteporfin photodynamic therapy at standard or reduced fluence level in patients with subfoveal CNV due to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients are men or women of age 50 or older.
* Patients have not received previous treatment for subfoveal choroidal neovascularization (CNV).
* Patients must have evidence of active or recurrent subfoveal CNV as confirmed by fluorescein angiography.
* The total lesion must be less than or equal to 9 disc areas in size, with a greatest linear distance of 5400 microns.
* Best corrected visual acuity, using ETDRS charts, of 20/40 to 20/320 (Snellen equivalent) in the study eye. Only one eye will assessed in the study.
* The CNV lesion must be primarily CNV (i.e. CNV equal to or greater than 50% of the lesion.
* The CNV is associated with only macular degeneration.
* Patient defers other approved treatments of subfoveal CNV associated with AMD.

Exclusion Criteria:

* Prior treatment for subfoveal choroidal neovascularization (CNV).
* Prior treatment for juxtafoveal or extrafoveal CNV involving previous antiangiogenic agent, photodynamic therapy, or intravitreal triamcinolone acetate.
* History of vitrectomy or submacular surgery in the study eye.
* Subretinal fibrosis accounting for more than 50% of the lesion.
* Non-CNV lesion components account for more than 50% of the total lesion components.
* CNV due to causes other than AMD.
* Retinal pigmented epithelial tear involving the center of the macula.
* Geographic atrophy involving the central macula.
* Any concurrent intraocular condition in the study eye that in the opinion of the investigator could require surgical or medical intervention during the course of the study (i.e. cataract).
* Active intraocular inflammation.
* Vitreous hemorrhage in the eye.
* History of spherical equivalent in the study eye greater than negative 8 diopters.
* Intraocular surgery within 2 months of study enrollment.
* Uncontrolled glaucoma in the study eye. Defined as intraocular pressure greater than 30mmHg despite treatment with anti-glaucoma medication.
* History of other disease, such as recent myocardial infarction, recent cerebral vascular accident, or uncontrolled hypertension that in the opinion of the investigator might render the subject at high risk for complication.
* Inability to comply with study or follow-up procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dante J Pieramici, MD, Principal Investigator — California Retina Consultants
Locations (2):
- United States (2):
  - California Retina Consultants, Bakersfield, California
  - California Retina Consultants, Santa Barbara, California

REFERENCES:
- See also: California Retina Consultants Website — http://www.californiaretina.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced Fluence: Reduced Fluence
  Bevacizumab and verteporfin photodynamic therapy: Patients will receive combination verteporfin with photodynamic therapy at reduced fluence [300mw/cm2] followed by intravitreal bevacizumab (1.25mg) on same day following photodynamic therapy.
- Standard Fluence: Standard Fluence
  Bevacizumab and visudyne photodynamic therapy: Patients will receive combination verteporfin photodynamic therapy with stand fluence [600mW/cm2] followed by intravitreal bevacizumab (1.25 mg) on the same day after photodynamic therapy.
Period: Overall Study
Arm/Group | Reduced Fluence | Standard Fluence
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Fluence | Standard Fluence | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Full Range); unit: years] | 79.0 [73 to 84] | 83.8 [75 to 94] | 81.4 [73 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22
visual acuity [Mean (Standard Deviation); unit: ETDRS letters] | 54.18 (13.7) | 60.5 (7.9) | 57.34 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity: Percentage of Patients Losing 3 or More Lines(15 Letters) of Visual Acuity From Baseline.
Time Frame: 1 Year
Measure: Number; unit: percent of participants
Arm/Group | Reduced Fluence | Standard Fluence
Number analyzed (Participants) | 11 | 11
percent of participants | 80 | 90

ADVERSE EVENTS:
Arm/Group | Reduced Fluence | Standard Fluence
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes